CLINICAL TRIAL: NCT04301570
Title: Validation Sonic Bone's Ultrasound System for Bone Age Assessment (BAUS)
Brief Title: Validation Sonic Bone's Ultrasound System for Bone Age Assessment
Acronym: BAUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Swiss Federal Institute of Sport Magglingen (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019-00526
Record Dates: First submitted 2020-03-05; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Bone Age Assessment
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound (Other): The intervention measurement is the determination of bone age using the ultrasound device.
  Interventions: Device: Ultrasound device
- XR (Other): The control measurement is the determination of the bone age by the imaging method using X-rays.
  Interventions: Radiation: XR

INTERVENTIONS:
Device: Ultrasound device — The measurement of bone age is performed via ultrasound with the "Ultrasound System for Bone Age Assessment (BAUS)" from Sonic Bone (SonicBone Medical Ltd., Rishon Lezion, Israel).
  Arms: Ultrasound
Radiation: XR — The measurement of bone age is performed via imaging procedure via X-ray (Röntgengerät, Stadler SE 4600, Littau, CH) of the left hand.
  Arms: XR

SUMMARY:
The selection of talents in junior sports is strongly influenced by the current physical conditions of the athletes. However, the physical abilities, for example in junior football, are largely dependent on the maturation and show a high degree of variability during puberty. For example, the maturity status in an U14 football team fluctuates by up to 5 years between early and late developed players. It is necessary to include the maturation in junior sports in selections in order to give all athletes the same chance of selection regardless of their maturity status. This will make selections fairer and the promotion of athletes with the highest potential will be better implemented. Bone age is considered to be an objective indicator of the maturation. For this purpose, a practicable and preferably radiation-free method for determining bone age is needed. A new medical device promises to determine bone age based on ultrasound technology. This now offers the chance to switch to a significantly less stressful technique. The aim of the study is to determine the quality criteria (validity and reliability) of this new method in order to decide whether the current gold standard of the X-ray method could be replaced by a less stressful method.

ELIGIBILITY:
Inclusion Criteria:

* Age between 10-18
* healthy
* voluntary participation
* consent of the participant or legal representative to participate in the project
* active in a sports club

Exclusion Criteria:

* pregnancy

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 416 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Bone Age Assessment using Ultrasound | 20 minutes
  The bone age is determined by the use of the new medical device according to the instructions for use.
Bone Age Assessment by imaging method using X-Ray | 20 minutes
  The gold standard is the determination of bone age according to the Tanner & Whitehouse (TW2) method using an X-ray image of the hand bone and subsequent calculation based on standardized comparison images (Tanner et al., 1975).

CONTACTS AND LOCATIONS:
Overall Officials: Jon Wehrlin, Dr. scient., Principal Investigator — Responsible for R+D
Locations (1):
- Swiss Federal Instistiution of Sport, Magglingen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malina RM, Cumming SP, Kontos AP, Eisenmann JC, Ribeiro B, Aroso J. Maturity-associated variation in sport-specific skills of youth soccer players aged 13-15 years. J Sports Sci. 2005 May;23(5):515-22. doi: 10.1080/02640410410001729928. PMID 16194999
- [Background] Malina RM, Rogol AD, Cumming SP, Coelho e Silva MJ, Figueiredo AJ. Biological maturation of youth athletes: assessment and implications. Br J Sports Med. 2015 Jul;49(13):852-9. doi: 10.1136/bjsports-2015-094623. PMID 26084525
- [Background] Malina RM, Coelho E Silva MJ, Figueiredo AJ, Carling C, Beunen GP. Interrelationships among invasive and non-invasive indicators of biological maturation in adolescent male soccer players. J Sports Sci. 2012;30(15):1705-17. doi: 10.1080/02640414.2011.639382. Epub 2012 Feb 3. PMID 22304621
- [Background] Tanner, J. M., Whitehouse, R., Cameron, N., Marshall, W., Healy, M., & Goldstein, H. (1975). Assessment of skeletal maturity and prediction of adult height (TW2 method) (Vol. 16): Academic Press London.